CLINICAL TRIAL: NCT03670147
Title: Effects of Paresthesia Free Spinal Cord Stimulation on Pain Intensity, Functional Improvement, Pain Thresholds and Sensory Perceptions in Chronic Pain Patients
Brief Title: Paresthesia Free Spinal Cord Stimulation (PF-SCS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit subjects due to Covid pandemic
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Shihab Ahmed, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018P-001645
Record Dates: First submitted 2018-08-01; First posted 2018-09-13 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: SCS; Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participant and study staff will be blinded. The study physicians will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Returns (Experimental): PF-SCS programming: in a blinded fashion, subjects will be asked to switch to the lowest amplitude program (LAP). Subjects whose pain returns after switching to the LAP will be considered Group 1.
  Interventions: Device: PF-SCS programming
- No Pain (Experimental): PF-SCS programming: in a blinded fashion, subjects will be asked to switch to the lowest amplitude program (LAP). Subjects whose pain does not return after switching to the LAP will be considered Group 2.
  Interventions: Device: PF-SCS programming

INTERVENTIONS:
Device: PF-SCS programming — In a blinded fashion, the study physician will ask subjects to switch their PF-SCS to the LAP.

SUMMARY:
The goal is to document efficacy of PF-SCS therapy in a blinded fashion and better understand how SCS therapy works in the clinical setting. Overall the investigators hope to improve patient care and selection of candidates who have the best potential for effective pain relief from an expensive and invasive therapy.

DETAILED DESCRIPTION:
The PF-SCS has 3 programs (P1, P2, P3) that can be used. At Visit 1, the study physician will review the PF-SCS program that the participant has been using. This program is known as the optimal program (OPP) and will be known as P1. The study physician will then designate the other two programs (P2 and P3); one of them will be identical to the OPP (P1) and the other program will be the LAP. The participant will be unaware if the LAP is assigned to P2 or P3. At the end of Visit 1, the study physician will have the participant switch from P1 to the LAP (P2 or P3). The participant will be reassured that if their pain returns after they switch programs, they can immediately call the study physician and will be switched back to the previous OPP (P1) without delay. The participants whose pain returns will be categorized as Group 1. The physician will document the time that had elapsed before their pain returned. This time will be considered as "carry over time" (COT) from PF-SCS. Only the study physicians will be aware of the programming parameters for P2 and P3. The rest of the study staff and participants will be blinded and will not be aware of the programming parameters for P2 and P3.

The participants whose pain remains stable while on the LAP will be categorized as Group 2. All participants will keep a daily diary for pain intensity, sleep and any other concerns that may arise related to the change of program.

At the end of Visit 1, a member of the study team will schedule Visit 2, between 14 to 28 days from Visit 1.

Phone call: A study physician will call subjects between 7-14 days after Visit 1. Group 1 participants will be asked to switch to the LAP (P2 or P3) before Visit 2. To minimize the duration of the LAP, Visit 2 will be scheduled within six hours from the end of COT. The Group 2 participants will attend Visit 2 without changing their LAP.

At Visit 2, participants will fill out questionnaires on pain intensity, sleep, activities and global impression. A blinded study staff will perform QST on the subject. At the end of Visit 2, Group 1 participants will be instructed to go back to the OPP (P1). At the end of Visit 2, Group 2 will be allowed to switch back to the OPP (P1).

The investigators will use quantitative sensory testing (QST) as a tool to objectively quantify the impact of SCS on heat pain threshold, heat pain tolerance and wind-up over the painful area and compare this with a non-painful area in each subject. QST will be performed at Visit 1 and Visit 2.

ELIGIBILITY:
Inclusion Criteria:

* Subject will be 18-80 years old
* Subject who is currently treated with PF-SCS (HF-10 or Burst-mode capable SCS system) for chronic pain

Exclusion Criteria:

* Subject has neurological disease or a condition causing chronic persistent sensory deficit to the painful area
* Those receiving remuneration for their pain treatment (pending litigation or ongoing litigation).
* Those unable to read English and complete the assessment instruments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
20% increase of NRS (numerical rating scale) pain scale | from date of consent until end of study (14-28 days)
  20% increase on low back pain NRS pain scale (0 = no pain and 10= maximum pain imaginable) while on LAP (lowest amplitude program) compared to OPP (optimal program).

SECONDARY OUTCOMES:
Quantitative Sensory Testing (QST) Results | from date of consent until end of study (14-28 days)
  Compare sensory perception on both the area of pain and the non-painful area on the opposite side while on the OPP (optimal program) and the LAP (lowest amplitude program). The following tests will be analyzed:
  * warm sensation (degrees Celsius)
  * heat pain threshold (degrees Celsius)
  * heat pain tolerance (degrees Celsius)
  * wind-up (NRS pain scale)
Daily diary results | from date of consent until end of study (14-28 days)
  Subject reported responses regarding their pain while using the OPP (optimal program):
  * global impression of change in pain (0=no pain, 10=worst pain)
  * impact on sleep and mood (0= does not interfere, 10= interferes completely)
  * daily living (0= does not interfere, 10= interferes completely)
  * enjoyment and general activity (0= does not interfere, 10= interferes completely)

CONTACTS AND LOCATIONS:
Overall Officials: Shihab Ahmed, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Center for Translational Pain Research, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No